CLINICAL TRIAL: NCT06376240
Title: The Effect of Pyridoxamine Supplementation on Microvascular Function in Type 2 Diabetes: a Double-blind Randomized Placebo-controlled Crossover Trial
Brief Title: The Effect of Pyridoxamine Supplementation on Microvascular Function in Type 2 Diabetes
Acronym: PYRAMID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Diabetes Fonds (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL85203.068.23
Record Dates: First submitted 2024-04-08; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes; Microvascular Function; Retinopathy, Diabetic; Nephropathy, Diabetic; Neuropathy, Diabetic
Keywords: Pyridoxamine; Advanced Glycation End Products; Methylglyoxal; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Retinopathy; Diabetic Nephropathies; Diabetic Neuropathies | interventions — Pyridoxamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment order AB (Experimental): Treatment with A (either pyridoxamine or placebo) in period 1 followed by treatment with B (either pyridoxamine or placebo) in period 2.
  Interventions: Dietary Supplement: Pyridoxamine 300mg per day; Other: Placebo 300mg placebo per day
- Treatment order BA (Experimental): Treatment with B (either pyridoxamine or placebo) in period 1 followed by treatment with A (either pyridoxamine or placebo) in period 2.
  Interventions: Dietary Supplement: Pyridoxamine 300mg per day; Other: Placebo 300mg placebo per day

INTERVENTIONS:
Dietary Supplement: Pyridoxamine 300mg per day — oral supplement
Other: Placebo 300mg placebo per day — oral supplement

SUMMARY:
Patients with type 2 diabetes have an increased risk of developing vascular complications. Microvascular dysfunction might be caused by the increased production of methylglyoxal under hyperglycaemic conditions. Methylglyoxal is a by-product of glycolysis and forms advanced glycation endproducts (AGEs) on proteins and DNA, thereby disrupting their function. Preventing methylglyoxal accumulation and AGEs formation may offer a therapeutic option for treating microvascular complications in diabetics. Pyridoxamine is a vitamin B6 vitamer that scavenges methylglyoxal and thereby inhibits the formation of AGEs. In this study, the researchers investigate whether pyridoxamine supplementation in type 2 diabetes improves microvascular function in the eye, kidney and skin, and reduces markers of endothelial dysfunction and glycation.

DETAILED DESCRIPTION:
Rationale:

People with diabetes have an increased risk of malfunctioning of the small blood vessels, e.g. in the eye and kidney, which can lead to blindness and kidney failure. These are serious complications, but to date there are no options to improve specifically the function of the small blood vessels. But why do people with diabetes have such an increased risk of dysfunction of the small blood vessels? The investigators have shown that a high glucose concentration in the blood plays an important role in the dysfunction of, particularly, the small blood vessels. A possible explanation for this dysfunction is an increased production of methylglyoxal, which arises from the breakdown of glucose. Methylglyoxal is a small but highly reactive molecule that can damage various organs and tissues. In several studies, the investigators found that methylglyoxal is increased in type 1 and type 2 diabetes and that methylglyoxal is associated with dysfunction of the smaller blood vessels. In our previous research in small laboratory animals, The investigators have shown that methylglyoxal directly causes damage of the small blood vessels. Because of these potentially harmful effects of methylglyoxal, the investigators have tried to reduce circulating methylglyoxal. In small laboratory animals, the investigators have found that the vitamin B6 isoform pyridoxamine inhibits the formation and accumulation of methylglyoxal, and improves vascular function. In a clinical trial in people with overweight, the investigators found that supplementation of pyridoxamine is safe and that methylglyoxal levels can be reduced, and the investigators found indications of an improvement of vascular function.

Objective:

Primary objective: to study whether pyridoxamine supplementation in type 2 diabetes improves microvascular function in the eye, kidney and skin, and reduces markers of endothelial dysfunction and glycation.

Secondary objective: to study whether pyridoxamine supplementation in type 2 diabetes improves glucose metabolism, advanced glycation endproduct (AGE) concentrations in blood plasma and skin, methylglyoxal, glyoxal and 3-deoxyglucose concentrations in blood plasma, adipokines and inflammatory markers in blood plasma, markers of dicarbonyl stress and oxidative stress in urine, liver fat, blood pressure, heart rate/ECG and body composition.

Study design:

The study will be conducted in a randomized, double blind, placebo-controlled manner. This intervention study includes two intervention periods of 8 weeks in a crossover design with a washout period of 4 weeks.

Study population:

Adult individuals (>18 years old) with type 2 diabetes, and with generalized microvascular dysfunction, i.e. an estimated glomerular filtration rate (eGFR) of 30-60 mL/min/1.73m2, and/or microalbuminuria of (albumin-creatinine ratio) 3-30 mg/mmol, and/or retinopathy (not proliferative), and/or neuropathy (any).

Intervention:

The daily dosage (300 mg) pyridoxamine or placebo will be supplied as three capsules of 100mg each per day, and are taken shortly before or during the meal.

Main study parameter:

The main study parameter is microvascular function in the eye, skin, plasma, and kidney measured by means of retinal funduscopy, adaptive optics funduscopy, optical coherence tomography (OCT), dynamic vessel analyser, skin laser doppler flowmetry, markers of endothelial function in the blood plasma, urinary albumin, and estimated glomerular filtration rate.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The number of measurements during each visit in this study is quite substantial. Nonetheless, the investigators expect that the burden for the subjects is limited since all measurements, except blood withdrawal, are non-invasive, and are performed while sitting or in a supine, relaxed, and comfortable position. Additionally, potential benefits of participating in this study are directly related to the possible beneficiary effects of pyridoxamine as showed in a previous clinical trial. Moreover, pyridoxamine supplementation in this previous clinical trial did not result in serious adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes,
* Generalized microvascular dysfunction, i.e.

  * eGFR 30-60 mL/min/1.73m2, and/or
  * Microalbuminuria albumin-creatinine ratio 3-30 mg/mmol, and/or
  * Retinopathy (not proliferative), and/or
  * Neuropathy (any).

Exclusion Criteria:

* Uncontrolled diabetes (i.e., hypoglycaemia >2 times/week and/or unstable HbA1c >9%),
* Use of >12 Units long-acting insulin per day,
* Use of short-acting insulin,
* Intraocular pressure ≥30 mmHg,
* History of glaucoma,
* Diagnosis of proliferative diabetic retinopathy,
* Diagnosis of diabetic macula edema,
* Albumine-creatinine ratio >30 mg/mmol,
* eGFR <30 mL/min/1.73m2,
* Diagnosis of epilepsy,
* Active cardiovascular disease,
* Alcohol usage >4 U/day,
* Drugs abuse,
* Use of systemic glucocorticosteroids,
* Higher grade hypertension
* Diagnosis of inflammatory disease,
* Use of an investigational product within the previous month,
* Unstable body weight,
* Pregnancy or lactation,
* Change in use of oral contraceptives or IUD,
* Unwillingness to give up being a blood donor (or having donated blood) from 8 weeks prior to the start of the study to end of study,
* Insufficient knowledge of the Dutch language,
* Inability to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Central retinal artery equivalent of the eye | 8 weeks
  in μm, measured with funduscopy

OTHER OUTCOMES:
eGFR | 8 weeks
  in ml/min/1.73m2
Microvascular function in skin | 8 weeks
  in %, measured with Laser Doppler Flowmetry
Markers of endothelial function and glycation in blood plasma. | 8 weeks
  in ng/ml, measured with ELISA, electrochemiluminicence technology and UPLC-MS/MS
Advanced glycation end products in skin | 8 weeks
  Measured with autofluorescent light
Advanced glycation end products in blood plasma and urine | 8 weeks
  in nmol/L, measured with UPLC-MS/MS
Adipokines and inflammatory markers in blood plasma | 8 weeks
  in mg/ml or pg/ml, measured with ELISA and electrochemiluminicence technology
Methylglyoxal, glyoxal and 3-deoxyglucose in blood plasma. | 8 weeks
  in nmol/L, measured with UPLC-MS/MS
Markers of dicarbonyl stress and oxidative stress in urine | 8 weeks
  in nmol/L, measured with UPLC-MS/MS
Glucose metabolism | 8 weeks
  Glucose iAUC, mmol/L x min, measured with Oral Glucose Tolerance Test
Liver fat | 8 weeks
  CAP score as measured with FibroScan
Systolic and diastolic blood pressure | 8 weeks
  in mmHg
Microvascular function eye | 8 weeks
  As measured with adaptive optics, optical coherence tomography angiography, and dynamic vessel analysis
Urinary albumin | 8 weeks
  in mg/24u

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Hospital Maastricht, Maastricht, Netherlands